CLINICAL TRIAL: NCT03302793
Title: Combined Peripheral (BreEStim) and Central Electrical Stimulation (tDCS) for Neuropathic Pain Management
Brief Title: Combined Peripheral (BreEStim) and Central Electrical Stimulation (tDCS) for Neuropathic Pain Management - Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sheng Li, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-14-0564 SCI
Record Dates: First submitted 2017-10-01; First posted 2017-10-05 (Actual); Results first posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- BreEStim and tDCS sham, then combined BreEStim and tDCS (Experimental): BreEStim is voluntary breathing controlled electrical stimulation.
  Interventions: Device: BreEStim; Device: tDCS; Device: tDCS sham
- Combined BreEStim and tDCS, then BreEStim and tDCS sham (Experimental): BreEStim is voluntary breathing controlled electrical stimulation. tDCS is transcranial direct current stimulation.
  Interventions: Device: BreEStim; Device: tDCS; Device: tDCS sham

INTERVENTIONS:
Device: BreEStim — BreEStim will applied for 10 to 20 minutes.
Device: tDCS — tDCS will be applied for 20 minutes.
Device: tDCS sham

SUMMARY:
This study looks at the effect of combined breathing-controlled electrical stimulation (BreEStim) and transcranial direct current stimulation (tDCS) on neuropathic pain after spinal cord injury, amputation, or brain injury. The hypothesis is that a single session of combined BreEStim and tDCS will produce an additive analgesic effect. This record covers the study in a population of spinal cord injury patients. Note that this study will also enroll healthy volunteers, brain injury patients, and amputation patients and that this study as applied to these other populations will be covered in separate ClinicalTrials.gov records.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 75 years
* male and female subjects
* has neuropathic pain after traumatic spinal cord injury
* has chronic pain, >3 months
* is stable on oral pain medications at least two weeks. (patients are allowed to continue their pain medications, i.e., no change in pain medications.)

Exclusion Criteria:

* currently adjusting oral pain medications for their neuropathic pain
* have pain, but not neuropathic (e.g., from inflammation at the incision wound of the residual limb or neuroma)
* have a pacemaker, or other metal and/or implanted devices
* have amputation in their arm(s)
* have spinal cord injury (SCI) involving impairment of arms
* have cognitive impairment from brain injury or are not able to follow commands, or to give consent
* have asthma or other pulmonary disease
* are not medically stable
* have preexisting psychiatric disorders
* alcohol or drug abuse
* have a history of seizures/Epilepsy, or taking benzodiazepines, anticonvulsants, and antidepressants.
* Mini-mental state examination (MMSE), a brief 30-point questionnaire test that is commonly used in the literature, will be used to screen for cognitive impairment. A brain injury patient with a score of 24 or lower on MMSE will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Li, MD, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- TIRR, Houston, Texas, United States

REFERENCES:
- [Result] Li S, Stampas A, Frontera J, Davis M, Li S. Combined transcranial direct current stimulation and breathing-controlled electrical stimulation for management of neuropathic pain after spinal cord injury. J Rehabil Med. 2018 Sep 28;50(9):814-820. doi: 10.2340/16501977-2379. PMID 30132010

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham tDCS and Then BreEStim; Then M1 tDCS and Then BreEstim; M1 tDCS and Then BreEStim; Then Sham tDCS and Then BreEstim: This study has a single-blinded, single-center, sham-controlled, crossover design. It included 2 separate visits, each with either a 20-min sham tDCS or M1 tDCS to the current dominant primary motor cortex(M1), both followed by a 20-min BreEStim to the median nerve(160 times) transcutaneously on the current dominant side.
Period: Overall Study
Arm/Group | Sham tDCS and Then BreEStim; Then M1 tDCS and Then BreEstim | M1 tDCS and Then BreEStim; Then Sham tDCS and Then BreEstim
Started | 6 | 6
Completed | 6 | 4
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: 2 subjects only finished Combined active tDCS (M1) and BreEStim section, but didn't attend the Sham tDCS and BreEStim section.
Groups:
- All Participants: This study has a single-blinded, single-center, sham-controlled, crossover design. It included 2 separate visits, each with either a 20-min sham tDCS or M1 tDCS to the current dominant primary motor cortex(M1), both followed by a 20-min BreEStim to the median nerve(160 times) transcutaneously on the current dominant side.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7
  Black | 2
  Hispanic | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Pain as Assessed by Visual Analogue Scale (VAS)
Description: A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. To allow a continuous assessment of pain, VAS uses a 10 cm line labelled at '0' with 'no pain' and '10' with 'worst pain'. The line is marked at a point corresponding to the assessment of the pain.
Time Frame: baseline, 10 minutes after tDCS, 10 minutes after BreEstim
Population: In the Sham tDCS and then BreEStim arm, only 10 participants were analyzed because 2 patients did not return for the second visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sham tDCS and Then BreEStim: This study has a single-blinded, single-center, sham-controlled, crossover design. It included a 20-min sham tDCS to the current dominant primary motor cortex(M1), followed by a 20-min BreEStim to the median nerve(160 times) transcutaneously on the current dominant side.
- Active tDCS (M1) and Then BreEStim: This study has a single-blinded, single-center, sham-controlled, crossover design. It included a 20-min active tDCS to the current dominant primary motor cortex(M1), followed by a 20-min BreEStim to the median nerve(160 times) transcutaneously on the current dominant side.
Arm/Group | Sham tDCS and Then BreEStim | Active tDCS (M1) and Then BreEStim
Number analyzed (Participants) | 10 | 12
units on a scale
  baseline | 6.0 (2.03) | 5.9 (1.65)
  After tDCS | 5.4 (2.26) | 5.3 (1.66)
  After BreEstim | 3.5 (1.91) | 3.1 (2.08)

2. Secondary Outcome: Electrical Pain Threshold
Description: Trimmed surface electrodes (1 inch by 1 inch) were used to examine electrical pain thresholds upon application of electrical stimulation (electrical stimulator 7SA, Digitimer). To measure electrical pain threshold, a pair of electrodes was placed next to each other centered on the thenar eminence (which is a group of muscles on the palm of the human hand at the base of the thumb); the intensity of electrical stimulation was started from the sensation threshold level (determined in outcome measure 3) and increased in steps of 1 mA; and subjects were instructed to close their eyes and to say ''yes'' when they first felt electrical stimulation painful. The electrical pain threshold is the mA level at which a participant first felt electrical stimulation painful. To improve consistency among subjects, they were advised that the pain threshold level was equivalent to 1 on the 0-10 VAS scale. Three repetitions were made and the average was used as the electrical pain threshold.
Time Frame: baseline, 10 minutes after tDCS, 10 minutes after BreEstim
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mA
Arm/Group | Sham tDCS and Then BreEStim | Active tDCS (M1) and Then BreEStim
Number analyzed (Participants) | 10 | 12
mA
  Baseline | 30.4 (25.53) | 35.0 (26.04)
  After tDCS | 31.1 (27.05) | 33.9 (26.37)
  After BreEstim | 34.5 (24.14) | 35.2 (21.58)

3. Secondary Outcome: Electrical Sensation Threshold
Description: Trimmed surface electrodes (1 inch by 1 inch) were used to examine electrical sensation threshold upon application of electrical stimulation (electrical stimulator 7SA, Digitimer). To measure electrical sensation threshold, a pair of electrodes was placed next to each other centered on the thenar eminence (which is a group of muscles on the palm of the human hand at the base of the thumb); the intensity of electrical stimulation was started from zero and gradually increased in steps of 0.1 mA; and subjects were instructed to close their eyes and to say ''yes'' when they explicitly felt electrical stimulation. The electrical sensation threshold is the mA level at which a participant explicitly felt electrical stimulation. Three repetitions were made and the average was used as the electrical sensation threshold.
Time Frame: baseline, 10 minutes after tDCS, 10 minutes after BreEstim
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mA
Arm/Group | Sham tDCS and Then BreEStim | Active tDCS (M1) and Then BreEStim
Number analyzed (Participants) | 10 | 12
mA
  Baseline | 7.3 (2.41) | 8.4 (2.59)
  After tDCS | 7.4 (2.84) | 8.1 (2.51)
  After BreEstim | 7.3 (2.66) | 8.3 (2.47)

ADVERSE EVENTS:
Time Frame: 16 hours after treatment
Arm/Group | Sham tDCS and Then BreEStim | Active tDCS (M1) and Then BreEStim
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 0/10 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-07): https://cdn.clinicaltrials.gov/large-docs/93/NCT03302793/Prot_SAP_000.pdf